CLINICAL TRIAL: NCT00976716
Title: An Open-Label, Multicenter Study To Evaluate The Efficacy, Safety And Tolerability Of Celecoxib (YM177) In Patients With Posttraumatic Pain
Brief Title: An Open-Label Study Of Celecoxib In Patients With Posttraumatic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3191357
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: posttraumatic pain
MeSH Terms: conditions — Pain | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celecoxib (Experimental)
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — Day 1
  * The first dose: Celecoxib 400mg
  * The second dose: Celecoxib 200mg during a period between 6 hours post-first dose and before bed
  Days 2 to 8 (Study drug should be taken until the dose scheduled after breakfast on the day of Day 8)
  - Celecoxib 200mg twice daily

SUMMARY:
To investigate efficacy, safety and tolerability of Celecoxib in patients with posttraumatic pain for the duration of 8 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with posttraumatic pain which is able to be controlled with an oral NSAID
* Patients with "pain" that meets both of the following criteria within 48 hours after injury:

"Pain" Pain intensity (Categorical): "Moderate pain" or "Severe pain" Pain intensity (VAS): 45.0 mm or more

* Patients with "inflammation" that meets the following criteria within 48 hours after injury.

"Inflammation" Categorical: "Mild", "Moderate" or "Severe"

Exclusion Criteria:

* Patients who have received analgesics and anaesthetics for injury
* Patients with a history/complication of aspirin-induced asthma
* Patients taking excluded medications
* Patients with a history/complication of ischaemic heart disease, serious cardiac arrhythmias, cardiac failure congestive and cerebrovascular disorder or with a history/plan of revascularization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Japan (11):
  - Pfizer Investigational Site, Funabashi, Chiba
  - Pfizer Investigational Site, Ichikawa, Chiba
  - Pfizer Investigational Site, Matsudo, Chiba
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Ageo, Saitama
  - Pfizer Investigational Site, Saitama-shi, Saitama
  - Pfizer Investigational Site, Edogawaku, Tokyo
  - Pfizer Investigational Site, Kotoku, Tokyo
  - Pfizer Investigational Site, Nerimaku, Tokyo
  - Pfizer Investigational Site, Toshimaku, Tokyo
  - Pfizer Investigational Site, Kofu, Yamanashi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191357&StudyName=An%20Open-Label%20Study%20Of%20Celecoxib%20In%20Patients%20With%20Posttraumatic%20Pain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 12 centers in Japan.
Groups:
- Celecoxib: Received the first dose of celecoxib 400 mg and the second dose of celecoxib 200 mg at least 6 hours apart on Day 1, followed by celecoxib 200 mg BID (twice daily) for up to 7 days from Day 2.
Period: Overall Study
Arm/Group | Celecoxib
Started | 80
Completed | 79
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib: Received the first dose of celecoxib 400 mg and the second dose of celecoxib 200 mg at least 6 hours apart on Day 1, followed by celecoxib 200 mg BID for up to 7 days from Day 2.
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.1 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 41

OUTCOME MEASURES:

1. Primary Outcome: Patient Impressions at Final Visit (the Number of Participants Who Have Rated "Excellent" and "Good")
Description: The patient impression of the study medication was entered in the patient diary based on the following categories: "excellent," "good," "fair" and "poor."
  Efficacy was based on the patient impression of the study medication ("excellent" and "good") from the first study medication until Final Visit.
Time Frame: 8 days
Population: The full analysis set (FAS) consisted of all patients who received at least one study medication and had at least one post-baseline efficacy endpoint measurement regardless of the primary or secondary endpoints. For the summary at Final Visit, the method of the last observation carried forward (LOCF) was used.
Measure: Number; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Participants | 70

2. Secondary Outcome: Patient Impressions Within 8 Days Post-first Dose (the Number of Subjects Who Have Rated "Excellent" and "Good")
Description: The patient impression of the study medication was entered in the patient diary based on the following categories: "excellent," "good," "fair" and "poor."
  Efficacy was based on the patient impression of the study medication ("excellent" and "good") from the first study medication until each time point.
Time Frame: 6 hours post first dose and before sleep on Day 1, before sleep on Day 2, Day 4 (Visit 2) and Day 8 (Visit 3)
Population: The FAS consisted of all patients who received at least one study medication and had at least one post-baseline efficacy endpoint measurement regardless of the primary or secondary endpoints.
Measure: Number; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Participants
  Day 1, 6 hours post first dose (n=80) | 44
  Day 1, before sleep (n=80) | 48
  Day 2, before sleep (n=80) | 55
  Visit 2 (Day 4), (n=80) | 60
  Visit 3 (Day 8), (n=68) | 60

3. Secondary Outcome: Pain Intensity (PI) of Pain at Rest (Spontaneous Pain) as Measured by Visual Analog Scale (VAS) Within 8 Days Post-first Dose
Description: The PI of pain at rest (spontaneous pain) was recorded on the 100 mm VAS in the patient diary, where 0 mm=no pain, 100 mm=worst possible pain.
Time Frame: Baseline, 2, 4 and 6 hours post first dose, and before sleep on Day 1, on awakening and before sleep on Days 2 to 7, on awakening on Day 8 and Visit 3 (Day 8)
Population: The FAS consisted of all patients who received at least one study medication and had at least one post-baseline efficacy endpoint measurement regardless of the primary or secondary endpoints. For the summary at Final Visit, the method of the LOCF was used.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
mm
  Baseline (n=80) | 59.9 (11.4)
  Day 1, 2 hours post first dose (n=80) | 47.3 (19.5)
  Day 1, 4 hours post first dose (n=80) | 42.5 (20.5)
  Day 1, 6 hours post first dose (n=80) | 40.3 (20.9)
  Day 1, before sleep (n=80) | 38.1 (20.0)
  Day 2, on awakening (n=80) | 34.8 (21.5)
  Day 2, before sleep (n=80) | 29.0 (22.0)
  Day 3, on awakening (n=80) | 24.8 (20.0)
  Day 3, before sleep (n=78) | 21.8 (19.1)
  Day 4, on awakening (n=78) | 18.4 (19.6)
  Day 4, before sleep (n=73) | 17.8 (18.9)
  Day 5, on awakening (n=73) | 15.3 (18.0)
  Day 5, before sleep (n=68) | 15.0 (18.7)
  Day 6, on awakening (n=68) | 12.4 (17.2)
  Day 6, before sleep (n=68) | 11.6 (17.3)
  Day 7, on awakening (n=68) | 11.3 (18.1)
  Day 7, before sleep (n=55) | 9.7 (16.2)
  Day 8, on awakening (n=55) | 8.6 (13.3)
  Visit 3 (Day 8) (n=73) | 7.2 (13.0)
  Final Visit (LOCF, n=80) | 7.3 (13.4)

4. Secondary Outcome: PI of Pain on Active Movement as Measured by VAS Within 8 Days Post-first Dose
Description: The PI of pain on active movement was recorded on the 100 mm VAS in the patient diary, where 0 mm=no pain, 100 mm=worst possible pain.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib
Number analyzed (Participants) | 79
mm
  Baseline (n=79) | 75.5 (12.7)
  Day 1, 2 hours post first dose (n=77) | 61.4 (20.2)
  Day 1, 4 hours post first dose (n=77) | 55.3 (21.0)
  Day 1, 6 hours post first dose (n=77) | 51.5 (20.6)
  Day 1, before sleep (n=77) | 49.3 (21.0)
  Day 2, on awakening (n=77) | 45.5 (21.4)
  Day 2, before sleep (n=77) | 39.7 (22.6)
  Day 3, on awakening (n=77) | 35.5 (22.3)
  Day 3, before sleep (n=75) | 32.4 (21.8)
  Day 4, on awakening (n=75) | 27.2 (22.9)
  Day 4, before sleep (n=70) | 26.4 (21.0)
  Day 5, on awakening (n=70) | 23.5 (21.4)
  Day 5, before sleep (n=66) | 23.2 (22.0)
  Day 6, on awakening (n=66) | 19.2 (20.4)
  Day 6, before sleep (n=66) | 18.2 (20.1)
  Day 7, on awakening (n=66) | 17.1 (21.7)
  Day 7, before sleep (n=55) | 15.5 (20.7)
  Day 8, on awakening (n=55) | 14.3 (20.0)
  Visit 3 (Day8) (n=71) | 12.1 (18.7)
  Final Visit (LOCF, n=78) | 11.8 (18.7)

5. Secondary Outcome: Pain Intensity Differences (PID) in Pain at Rest (Spontaneous Pain) Within 8 Days Post-first Dose
Description: The PID score was obtained by subtracting the PI (by VAS: 0 mm=no pain, 100 mm=worst possible pain) at each time point from the Baseline PI score. Increase in PID scores indicated a lessening of subjects' pain compared to baseline scores; higher scores indicated a greater reduction in pain.
Time Frame: Two, 4 and 6 hours post first dose, and before sleep on Day 1, on awakening and before sleep on Days 2 to 7, on awakening on Day 8 and Visit 3 (Day 8)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
mm
  Day 1, 2 hours post first dose (n=80) | 12.6 (14.8)
  Day 1, 4 hours post first dose (n=80) | 17.4 (16.0)
  Day 1, 6 hours post first dose (n=80) | 19.6 (16.3)
  Day 1, before sleep (n=80) | 21.8 (16.8)
  Day 2, on awakening (n=80) | 25.1 (19.1)
  Day 2, before sleep (n=80) | 30.9 (20.8)
  Day 3, on awakening (n=80) | 35.1 (18.7)
  Day 3, before sleep (n=78) | 37.9 (18.8)
  Day 4, on awakening (n=78) | 41.3 (19.7)
  Day 4, before sleep (n=73) | 41.8 (19.2)
  Day 5, on awakening (n=73) | 44.3 (18.4)
  Day 5, before sleep (n=68) | 45.4 (19.5)
  Day 6, on awakening (n=68) | 48.0 (17.7)
  Day 6, before sleep (n=68) | 48.8 (18.1)
  Day 7, on awakening (n=68) | 49.2 (19.0)
  Day 7, before sleep (n=55) | 50.2 (18.7)
  Day 8, on awakening (n=55) | 51.3 (17.3)
  Visit 3 (Day 8) (n=73) | 52.4 (15.5)
  Final Visit (LOCF, n=80) | 52.6 (15.2)

6. Secondary Outcome: PID in Pain on Active Movement Within 8 Days Post-first Dose
Description: The PID score was obtained by subtracting the PI at each time point from the Baseline PI score. Increase in scores indicated a lessening of subjects' pain compared to baseline scores; higher scores indicated a greater reduction in pain.
Time Frame: 2, 4 and 6 hours post first dose, and before sleep on Day 1, on awakening and before sleep on Days 2 to 7, on awakening on Day 8 and Visit 3 (Day 8)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Celecoxib
Number analyzed (Participants) | 79
mm
  Day 1, 2 hours post first dose (n=77) | 14.3 (16.6)
  Day 1, 4 hours post first dose (n=77) | 20.4 (17.1)
  Day 1, 6 hours post first dose (n=77) | 24.3 (17.5)
  Day 1, before sleep (n=77) | 26.5 (17.5)
  Day 2, on awakening (n=77) | 30.3 (19.2)
  Day 2, before sleep (n=77) | 36.1 (22.0)
  Day 3, on awakening (n=77) | 40.2 (21.2)
  Day 3, before sleep (n=75) | 43.2 (21.5)
  Day 4, on awakening (n=75) | 48.5 (22.3)
  Day 4, before sleep (n=70) | 49.5 (20.6)
  Day 5, on awakening (n=70) | 52.5 (20.8)
  Day 5, before sleep (n=66) | 53.5 (21.6)
  Day 6, on awakening (n=66) | 57.5 (19.7)
  Day 6, before sleep (n=66) | 58.4 (19.9)
  Day 7, on awakening (n=66) | 59.6 (21.4)
  Day 7, before sleep (n=55) | 62.1 (20.6)
  Day 8, on awakening (n=55) | 63.3 (20.6)
  Visit 3 (Day 8) (n=71) | 63.6 (18.6)
  Final Visit (LOCF, n=78) | 63.7 (18.1)

7. Secondary Outcome: Sum of Pain Intensity Differences (SPID) for Pain at Rest (Spontaneous Pain) and on Active Movement Until 6 Hours Post-first Dose
Description: The SPID was derived according to the following rule: each PID was weighted by the width of time interval between previous and current time points in hours and summed up to 6 hours post-first dose
Time Frame: 6 hours
Population: The FAS consisted of all patients who received at least one study medication and had at least one post-baseline efficacy endpoint measurement. If a patient withdrew the study before 6 hours on Day 1 and the measurement of the PI at 6 hours on Day 1 was missing, the LOCF method was used for the PI at 6 hours on Day 1 to derive the SPID.
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
mm
  Pain at rest (n=80) | 99.3 [79.9 to 118.7]
  Pain on active movement (n=77) | 118.2 [96.7 to 139.6]

8. Secondary Outcome: Peak Pain Intensity Difference (PPID) for Pain at Rest (Spontaneous Pain) and on Active Movement Until 6 Hours Post-first Dose
Description: The PPID was obtained by subtracting the maximum value of pain intensity (PI) at a time point among 2 to 6 hours post first dose from baseline value of PI for each patient.
Time Frame: Two, 4 and 6 hours post first dose
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
mm
  Pain at rest (n=80) | 22.2 [18.6 to 25.8]
  Pain on active movement (n=77) | 26.7 [22.6 to 30.7]

9. Secondary Outcome: Severity of Inflammatory Symptoms (Swelling) Within 8 Days Post-first Dose
Description: The investigator assessed the swelling, using the categories "None," "Mild," "Moderate," and "Severe" at Baseline, Visit 2 (Day 4), Visit 3 (Day 8) and Final Visit.
Time Frame: Baseline, Days 4 (Visit 2) and 8 (Visit 3)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Participants
  None at Baseline (n=80) | 0
  None at Visit 2 (Day 4) (n=80) | 5
  None at Visit 3 (Day 8) (n=68) | 38
  None at Final Visit (n=80) | 41
  Mild at Baseline (n=80) | 24
  Mild at Visit 2 (Day 4) (n=80) | 69
  Mild at Visit 3 (Day 8) (n=68) | 26
  Mild at Final Visit (n=80) | 35
  Moderate at Baseline (n=80) | 48
  Moderate at Visit 2 (Day 4) (n=80) | 5
  Moderate at Visit 3 (Day 8) (n=68) | 4
  Moderate at Final Visit (n=80) | 4
  Severe at Baseline (n=80) | 8
  Severe at Visit 2 (Day 4) (n=80) | 1
  Severe at Visit 3 (Day 8) (n=68) | 0
  Severe at Final Visit (n=80) | 0

10. Secondary Outcome: Severity of Inflammatory Symptoms (Redness) Within 8 Days Post-first Dose
Description: The investigator assessed the redness, using the categories "None," "Mild," "Moderate," and "Severe" at Baseline, Visit 2 (Day 4), Visit 3 (Day 8) and Final Visit.
Time Frame: Baseline, Days 4 (Visit 2) and 8 (Visit 3)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Participants
  None at Baseline (n=80) | 16
  None at Visit 2 (Day 4) (n=80) | 51
  None at Visit 3 (Day 8) (n=68) | 64
  None at Final Visit (n=80) | 73
  Mild at Baseline (n=80) | 40
  Mild at Visit 2 (Day 4) (n=80) | 28
  Mild at Visit 3 (Day 8) (n=68) | 4
  Mild at Final Visit (n=80) | 7
  Moderate at Baseline (n=80) | 19
  Moderate at Visit 2 (Day 4) (n=80) | 1
  Moderate at Visit 3 (Day 8) (n=68) | 0
  Moderate at Final Visit (n=80) | 0
  Severe at Baseline (n=80) | 5
  Severe at Visit 2 (Day 4) (n=80) | 0
  Severe at Visit 3 (Day 8) (n=68) | 0
  Severe at Final Visit (n=80) | 0

11. Secondary Outcome: Severity of Inflammatory Symptoms (Localized Warmth) Within 8 Days Post First Dose
Description: The investigator assessed the localized warmth, using the categories "None," "Mild," "Moderate," and "Severe" at Baseline, Visit 2 (Day 4), Visit 3 (Day 8) and Final Visit.
Time Frame: Baseline, Days 4 (Visit 2) and 8 (Visit 3)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Participants
  None at Baseine (n=80) | 8
  None at Visit 2 (Day 4) (n=80) | 63
  None at Visit 3 (Day 8) (n=68) | 66
  None at Final Visit (n=80) | 76
  Mild at Baseine (n=80) | 43
  Mild at Visit 2 (Day 4) (n=80) | 17
  Mild at Visit 3 (Day 8) (n=68) | 2
  Mild at Final Visit (n=80) | 4
  Moderate at Baseine (n=80) | 23
  Moderate at Visit 2 (Day 4) (n=80) | 0
  Moderate at Visit 3 (Day 8) (n=68) | 0
  Moderate at Final Visit (n=80) | 0
  Severe at Baseine (n=80) | 6
  Severe at Visit 2 (Day 4) (n=80) | 0
  Severe at Visit 3 (Day 8) (n=68) | 0
  Severe at Final Visit (n=80) | 0

12. Secondary Outcome: Withdrawal Due to Lack of Efficacy
Description: The number of subjects who withdrew due to insufficient clinical response was evaluated.
Time Frame: 8 days
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Participants | 0

13. Secondary Outcome: Summary of Adverse Events
Description: The number of subjects who experienced adverse events (AEs; all-causality and treatment-related) based on safety assessment was summarized. The severity and seriousness of treatment-emergent AEs as well as discontinuations, dose reductions and temporary discontinuations (DR/TD) due to treatment-emergent AEs were also summarized.
Time Frame: 8 days
Population: The safety analysis set consisted of all patients who had taken at least one study medication.
Measure: Number; unit: Participants
Arm/Group | Celecoxib
Number analyzed (Participants) | 80
Participants
  AEs: all-causality | 10
  AEs: treatment-related | 8
  Severe AEs: all-causality | 0
  Severe AEs: treatment-realted | 0
  Serious AEs: all-causality | 0
  Serious AEs: treatment-related | 0
  Discontinuation due to all-causality AEs | 1
  Discontinuation due to treatment-related AEs | 1
  DR/TD due to all-causality AEs | 0
  DR/TD due to treatment-related AEs | 0

ADVERSE EVENTS:
Time Frame: 8 days
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 10/80
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=80)
Diarrhoea (Gastrointestinal disorders) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Beta 2 microglobulin urine increased (Investigations) | 5
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 2
Urobilin urine present (Investigations) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.